CLINICAL TRIAL: NCT06870227
Title: Effect of Scenario-Based Simulation on Clinical Learning, Confidence and Satisfaction of Midwifery Students in Management of Eclampsia Crisis in Labor
Brief Title: Scenario-Based Simulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Ph.D., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024/572
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Simulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Reality Simulator (Experimental): Eclampsia Crisis in Labor management training will be given by the responsible investigator, and then one of the groups will be allocated by randomization. Using High Reality Simulator will perform emergency Eclampsia Crisis in Labor. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one.
  Interventions: Other: Using High Reality Simulator
- control group (No Intervention): Using model will perform emergency y Eclampsia Crisis in Labor. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one.

INTERVENTIONS:
Other: Using High Reality Simulator — Using High Reality Simulator will perform emergency eclampsia in labour
  Arms: High Reality Simulator

SUMMARY:
The aim of this study is to determine the effect of Scenario-Based Simulation on Clinical Learning, Confidence and Satisfaction of Midwifery Students in Management of Eclampsia Crisis in Labor

DETAILED DESCRIPTION:
Hypotheses 01; there was no difference between the clinical learning score of the experimental group and the pain score of the control group.

H02; there was no difference between the confidence score of the experimental group and the confidence score of the control group.

H03; there was no difference between the satisfaction score of the of the experimental group and the satisfaction score of the control group.

The study will be carried out in two different groups. The practice will start with meeting the students. After the students are evaluated in terms of eligibility criteria for the research, the students who are eligible will be informed about the research and written informed consent will be obtained from the students who accept. The random distribution of students to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Eclampsia Crisis in Labor training will be given by the responsible investigator, and then one of the groups separated by randomization will perform Eclampsia Crisis in Labor first care on the second group model using High Reality Simulator. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Take the Obstetric Emergencies course

Exclusion Criteria:

* Not volunteering to participate in the study
* Not taking the obstetric emergencies course

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-Confidence/Competence in Patient Intervention Scale | immediately after intervention
  The validity and reliability study of the scale was conducted by Terzioğlu et al (2012). The scale was developed for health professional students who had experience in teaching based on scenario-based simulation. 3 factors were obtained in the explanatory factor analysis. The three factors were classified as clinical practice (11 items), psychological support (4 items) and health care system knowledge (3 items). The validity results of the scale were evaluated between 0.80 and 0.94. The Cronbach Alpha internal consistency coefficient of the scale was 0.947. The scale contains a total of 18 items and is evaluated according to the 5-point Likert system.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)